CLINICAL TRIAL: NCT06961695
Title: Assessing the Effectiveness of a Mindfulness-Based Virtual Reality Intervention to Reduce Pain in Postoperative Patients: A Controlled Clinical Study
Brief Title: The Efficacy of a Mindfulness-Based Virtual Reality Intervention to Reduce Pain in Postoperative Patients
Acronym: VR-MindPain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Cluj-Napoca County Emergency Clinical Hospital, Surgery Department 2 (Unknown)
Responsible Party: Principal Investigator, Roxana Cardos, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6997/27.02.2025
Record Dates: First submitted 2025-04-16; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Anxiety Preoperative
Keywords: Postoperative Pain; Mindfulness-Based Intervention; Pain Management; Chronic Pain Prevention; Virtual Reality
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR Mindfulness Intervention Group (Experimental): Participants in this arm will undergo a structured protocol including a VR-based mindfulness intervention. Patients are guided through psychoeducation about mindfulness, and the VR procedure. Patients are invited to express their worries about the intervention or the surgery, which are normalized and addressed through reflective listening. The mindfulness session in VR lasts approximately 10 minutes and is supervised by the clinical psychologist.
  A structured debriefing follows the VR session, using the 4Fs model:
  Feelings: How did the patient feel during the session? Findings: Did they discover anything helpful or meaningful? Futures: How can they apply mindfulness during hospitalization or at home? Follow-up: They receive a home practice suggestion (4x4 breathing technique) connected to a meaningful thought, image, or feeling from the VR session.
  Assesments at four time points.
  Interventions: Behavioral: VR Mindfulness-Based Relaxation
- Treatment as Usual (TAU) Group (No Intervention): Participants in this group will receive the standard preoperative and postoperative care provided by the hospital, without any additional intervention from the research team.
  Assesments at 3 time points.
  1. Before the intervention (Day 1)
  2. After surgery (Day 2)
  3. Two weeks after surgery (follow-up)

INTERVENTIONS:
Behavioral: VR Mindfulness-Based Relaxation — VR Mindfulness-Based Relaxation is a behavioral intervention that utilizes a VR application designed to reduce anxiety and promote relaxation. Participants in the experimental group will undergo a single VR session, scheduled on the day of hospital admission (one day prior to surgery).
  The session lasts approximately 10 minutes and features an immersive beach environment combined with an audio-guided mindfulness exercise focused on breath awareness. Following the session, participants will engage in a brief, structured debriefing, during which they will reflect on what they felt, what they discovered, and how they can apply these insights during their hospital stay.
  Participants will also be instructed to practice the 4-1-4 breathing technique three times per day during hospitalization. This technique involves inhaling for 4 seconds, holding the breath for 1 second, and exhaling for 4 seconds. It is intended to promote relaxation and support autonomic nervous system regulation.
  Arms: VR Mindfulness Intervention Group

SUMMARY:
The goal of this randomized clinical trial is to evaluate whether a virtual reality (VR) mindfulness intervention can reduce anxiety and postoperative pain in adults undergoing surgery, primarily hernia and varicose vein procedures.

The main research questions are:

* Does a preoperative VR mindfulness intervention reduce anxiety before surgery?
* Does this reduction in anxiety result in lower postoperative pain compared to usual care?
* Does the intervention help prevent chronic pain two weeks after surgery? Researchers will compare a VR mindfulness intervention group with a treatment-as-usual (TAU) group to assess the intervention's effectiveness.

Participants will:

* Be randomly assigned to one of two groups:

  * Experimental group: Receive a VR mindfulness session on the first day of hospitalization (one day before surgery).
  * Control group: Receive standard hospital care (no intervention).
* Complete psychological and pain assessments at four time points:

  1. Before the intervention (Day 1)
  2. Immediately after the intervention (only the experimental group, Day 1)
  3. After surgery (Day 2)
  4. Two weeks after surgery (follow-up)
* Report pain intensity using the Numeric Rating Scale (NRS) at four postoperative time points.

Before enrollment, participants will undergo a structured interview to assess eligibility.

This study aims to determine whether reducing preoperative anxiety through VR mindfulness contributes to improved pain management and a lower risk of developing chronic pain following surgery.

DETAILED DESCRIPTION:
Study Objective:

This study aims to assess the efficacy of a virtual reality (VR)-based mindfulness relaxation intervention in reducing preoperative anxiety, postoperative pain, and the risk of chronic pain two weeks after surgery.

Study Design:

This is a randomized controlled trial (RCT) comparing two groups:

1. Experimental Group - Participants will receive a VR mindfulness-based relaxation intervention prior to surgery.
2. Control Group - Participants will receive treatment as usual (TAU), with no additional intervention.

Intervention:

The VR mindfulness-based relaxation program will be administered on the day of hospitalization, one day prior to surgery.

The session will last 10-15 minutes and includes:

* A guided mindfulness exercise focused on breath awareness and relaxation.
* A virtual beach environment designed to enhance calm and reduce anxiety.
* A brief debriefing session following the second VR exposure (if applicable).

Assessments and Outcome Measures:

Structured psychological and pain assessments will be conducted at four time points:

1. Before the intervention (Day 1)
2. Immediately after the intervention (Day 1)
3. After surgery (Day 2)
4. Two weeks after surgery (follow-up)

Data Analysis:

* A Multivariate Analysis of Variance (MANOVA) with a mixed design (within-between interaction) will be used to assess differences across multiple dependent variables.
* Repeated measures MANOVA will be applied to examine longitudinal changes and interactions between time and group.

Expected Impact:

This study seeks to determine whether reducing preoperative anxiety through a VR mindfulness intervention improves postoperative pain management and reduces the likelihood of developing chronic pain. If effective, the intervention could be integrated into routine preoperative care protocols to enhance patient outcomes and overall recovery experiences.

ELIGIBILITY:
Inclusion Criteria

* The participant is scheduled for surgery and is currently hospitalized for hernia or varicose vein procedures.
* The participant is on the hospital's surgical waiting list.
* The participant is willing and able to provide informed consent.
* The participant agrees to participate in the study and to complete all required assessments during hospitalization and at follow-up (either at home or during post-operative medical visits).

Exclusion Criteria

* Inability to provide informed consent due to mental incompetence (e.g., intellectual disability, dementia); mild cognitive impairment does not constitute an exclusion criterion.
* Limited proficiency in the Romanian language.
* Active substance use or alcohol use disorders that, in the opinion of the investigators, may interfere with participation.
* History of motion sickness.
* Severe visual impairment (e.g., inability to see clearly without glasses); patients who use contact lenses are not excluded.
* Use of strong opioids (e.g., morphine).
* Current suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Brief Pain Inventory (BPI) . | The BPI will be administered at three time points: preoperatively (Day 1 of hospitalization), postoperatively (Day 2, the day of surgery), and at follow-up (2 weeks after surgery).
  This tool assesses both pain intensity and its impact on daily functioning (e.g., sleep, work, social interactions). The BPI consists of 9 items, each rated on a 0-10 scale, where 0 indicates no pain or interference and 10 represents the worst possible pain or interference.
Change in Pain Intensity Measured by Numeric Rating Scale (NRS) | The NRS will be administered four times throughout the day following the surgery.
  Participants will rate their pain intensity on a 0-10 scale, where 0 indicates no pain and 10 represents the worst imaginable pain. NRS assessments will be conducted at four postoperative time points. This approach helps minimize the influence of analgesics and anesthetics on reported pain levels. By spreading out the measurements, we reduce the risk that a single time point reflects only the temporary effects of medication, thus allowing for more reliable and valid comparisons between treatment groups.

SECONDARY OUTCOMES:
Change in Anxiety Levels Measured by State-Trait Anxiety Inventory - State version (STAI-S) | STAI-S measures will be administered: Preoperative/Pre-intervention (Day 1 of hospitalization) Post-intervention (Day 1, within 15 minutes after the VR session), Postoperative (Day 2, day of surgery), Follow-up (2 weeks after surgery).
  State-Trait Anxiety Inventory - state version (STAI-S) Measures state anxiety (how the participant feels "at this moment"). Contains 20 items rated on a 4-point Likert scale (from "Not at all" to "Very much").
  The scores range between 20 (no anxiety) and 80 (high anxiety)
Change in Anxiety Levels Measured by State-Trait Anxiety Inventory - Trait version (STAI-T) | STAI-T will be administered preoperatively, on Day 1 of hospitalization.
  The STAI-T measures trait anxiety, referring to how the participant generally feels. It consists of 20 items rated on a 4-point Likert scale, ranging from "Almost never" to "Almost always." Total scores range from 20 to 80, with higher scores indicating greater levels of anxiety.
Change in Anxiety Levels Measured by Hospital Anxiety and Depression Scale (HADS). | Preoperative/Pre-intervention (Day 1 of hospitalization) Postoperative (Day 2, day of surgery) Follow-up (2 weeks after surgery)
  Hospital Anxiety and Depression Scale (HADS):
  Evaluates anxiety and depression symptoms in hospitalized patients. Consists of 14 items divided into two subscales (anxiety and depression), each rated from 0 (absent) to 3 (severe).
  Total anxiety scores range from:
  0-7 (normal) 8-10 (borderline abnormal) 11-21 (abnormal)

OTHER OUTCOMES:
Change in Quality of Life Measured by EUROHIS-QOL. | Preoperative/Pre-intervention (Day 1 of hospitalization), Postoperative (Day 2, day of surgery), and Follow-up (2 weeks after surgery)
  Quality of life will be assessed using the EUROHIS-QOL 8-Item Index, a validated short-form version of the WHOQOL-BREF, designed for rapid assessment of subjective well-being.
  EUROHIS-QOL Scale Details:
  Consists of 8 items covering four key domains:
  Physical health (e.g., energy levels, ability to perform daily activities) Psychological well-being (e.g., satisfaction with life, emotional balance) Social relationships (e.g., satisfaction with personal relationships) Environment (e.g., financial security, living conditions)
  Each item is rated on a 5-point Likert scale, where higher scores indicate better quality of life.
Change in Sleep Quality Measured by Pittsburgh Sleep Quality Index (PSQI) | Preoperative/Pre-intervention (Day 1 of hospitalization), Postoperative (Day 2, day of surgery), and Follow-up (2 weeks after surgery)
  SQI Scale Details:
  Consists of 19 items grouped into 7 components: Subjective sleep quality, Sleep latency (time taken to fall asleep), Sleep duration, Sleep efficiency, Sleep disturbances, Use of sleep medication, Daytime dysfunction.
  Each component is scored from 0 to 3, where higher scores indicate greater sleep impairment.
  The total PSQI score ranges from 0 to 21, with a score ≥5 indicating poor sleep quality.
Change in Emotional Balance Measured by the Equanimity Scale-16 (ES-16) | Preoperative/Pre-intervention (Day 1 of hospitalization), Postoperative (Day 2, day of surgery), and Follow-up (2 weeks after surgery)
  Emotional balance will be assessed using the Equanimity Scale-16 (ES-16), a validated self-report instrument designed to measure the ability to accept internal experiences (thoughts, emotions, bodily sensations) without reacting impulsively.
  ES-16 Scale Details:
  Contains 16 items divided into two subscales:
  Experiential acceptance - Measures the ability to acknowledge and accept emotional experiences.
  Non-reactivity - Assesses the capacity to refrain from impulsive reactions to emotions.
  Each item is rated on a Likert scale from 1 (strongly disagree) to 5 (strongly agree).
  Higher scores indicate greater emotional balance and equanimity.
Change in Pain Catastrophizing Measured by the Pain Catastrophizing Scale (PCS) | Preoperative/Pre-intervention (Day 1 of hospitalization), Postoperative (Day 2, day of surgery), and Follow-up (2 weeks after surgery)
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), a self-report instrument designed to measure exaggerated negative responses to pain experiences.
  PCS Scale Details:
  Contains 13 items assessing three subdomains:
  Rumination - Persistent focus on pain-related thoughts. Magnification - Exaggeration of the perceived threat of pain. Helplessness - Feelings of being unable to manage pain. Items are rated on a Likert scale from 0 (never) to 4 (all the time). The total PCS score is obtained by summing individual item scores, with higher scores indicating greater pain catastrophizing.
Change in Mindful Attention and Awareness Measured by the Mindful Attention Awareness Scale (MAAS) | Immediately after the VR intervention (within 15 minutes).
  The Mindful Attention Awareness Scale (MAAS) is a validated instrument designed to assess individual differences in mindfulness, specifically the frequency of present-moment awareness and attention. It consists of 15 items, each rated on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never), with higher scores indicating greater mindfulness and present-moment awareness. Changes in MAAS scores will be analyzed to determine whether the VR mindfulness-based relaxation intervention enhances mindful awareness, potentially contributing to improved emotional regulation and pain perception.
Screening for Cognitive Function Measured by the Montreal Cognitive Assessment (MoCA) | Pre-intervention (Day 1 of hospitalization), if cognitive impairment is suspected based on clinical observation.
  Montreal Cognitive Assessment (MoCA) is a 30-point cognitive screening tool designed to detect mild cognitive impairment. The assessment evaluates multiple cognitive domains, including attention, concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The test comprises various tasks that collectively contribute to the total score of 30 points. Administration time is approximately 10 minutes, and a score of 26 or above is generally considered normal.
Presence Experience Measured by the Presence Questionnaire (PQ) | Immediately after the VR intervention (within 15 minutes).
  The Presence Questionnaire (PQ) is a validated instrument designed to assess the degree to which individuals feel immersed and engaged in a virtual environment. It evaluates multiple dimensions of presence, including involvement, sensory fidelity, adaptation/immersion, and interface quality. The questionnaire consists of 32 items rated on a 7-point Likert scale, with higher scores indicating a stronger sense of presence. This measure will be used to explore how engagement in the VR mindfulness relaxation intervention influences participants' perception of presence and its potential relationship with anxiety reduction, pain perception, and psychological well-being.
Simulator Sickness Symptoms Measured by Simulator Sickness Questionnaire (SSQ) | The SSQ will be administered immediately after the VR intervention (within 15 minutes)
  The Simulator Sickness Questionnaire (SSQ) consists of 16 symptoms grouped into three components: Nausea (e.g., increased salivation, stomach awareness), Oculomotor (e.g., eyestrain, blurred vision), and Disorientation (e.g., dizziness, vertigo). Each symptom is rated on a 4-point Likert scale ranging from 0 (none) to 3 (severe). Subscale scores and a total score are calculated using standardized weighting formulas, with higher scores indicating more severe symptoms of simulator sickness.